CLINICAL TRIAL: NCT05772611
Title: Characterization of Immune-response in Autoimmune Encephalitis and Paraneoplastic Neurological Syndromes
Acronym: Car-Te-Cell
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 788
Record Dates: First submitted 2023-02-14; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Autoimmune Encephalitis; Paraneoplastic Neurological Syndrome
Keywords: autoimmune encephalitis; paraneoplastic neurological syndromes; genetic
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Immunologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, DNA, cells, CSF collected at diagnosis time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Antibody characterized: Patients with well-characterized antibody (HU, YO, RI, CASPR2, NMDAr, GAD, …)
  Interventions: Biological: Genetic and immunology tests
- Atypical: Patients with atypical antibody
  Interventions: Biological: Genetic and immunology tests
- Without antibody: Patients without antibody
  Interventions: Biological: Genetic and immunology tests

INTERVENTIONS:
Biological: Genetic and immunology tests — This is a non-interventional study involving clinical data and biological samples (blood, DNA, CSF, cells). Clinical data are collected for the center and samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL) (including tissue, cells or biological fluids) and genetic analysis for research purposes.

SUMMARY:
Autoimmune encephalitis (AE) and paraneoplastic neurological syndromes (PNS) are rare neuroimmune syndromes with a wide range of clinical presentation but without pathognomonic clinical sign facilitating the diagnosis. A lot of differential diagnoses are possible such as neurodegenerative diseases or viral infections. Although rare the diagnosis of AE or PNS is essential because despite severe neurological symptoms, patients can be cured by appropriate immunotherapy. Autoantibodies highly specific of AE and PNS has been described in the serum and cerebrospinal fluid of the patients and can be used as biomarkers of the disease. Their presence can predict an autoimmune origin and in many cases a good prognosis after immunotherapy. However, if some autoantibodies are now well-characterized and industrial kits have been developed to detect them, in numerous cases of highly suspect AE or PNS no specific autoantibodies are identified leading frequently to an inappropriate treatment. Furthermore, as the mechanisms of AE and PNS is still unknown, treatments are not optimal and in some cases inefficient. There is no prognosis biomarker able to predict the patient's sensitivity to immunotherapy and there are only few clues to know how the immune system can provoke the neuropsychiatric symptoms observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with neurological disorder
* Patient with antibodies or not in sera or CSF

Exclusion Criteria:

- No available clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with auto-immune encephalitis suspected and antibody characterized or not.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between biological results and clinical data | Through study completion, an average of 1year
  This measure will compare the result of immunological and genetic makers with clinical data of each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France